CLINICAL TRIAL: NCT05002452
Title: Observational Study of Factors Predicting Therapeutic Effects and Clinical Prognosis After Hepatic Artery Infusion Chemotherapy (HAIC) for Locally Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Observational Study of Factors Predicting Therapeutic Effects and Clinical Prognosis After HAIC for Locally Advanced HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Professor, Sun Yat-sen University
Other Study IDs: B2021-107-01
Record Dates: First submitted 2021-08-07; First posted 2021-08-12 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Arterial infusion chemotherapy; FOLFOX
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Locally Advanced HCC Patients: Patients which are diagnosed with locally advanced hepatocellular carcinoma (HCC) will receive standard HAIC treatment.
  Interventions: Other: Search of factors predicting therapeutic effects and prognosis

INTERVENTIONS:
Other: Search of factors predicting therapeutic effects and prognosis — There factors are collected in preoperative routine blood examination, preoperative radiological imaging and pathological examination.

SUMMARY:
Prospective single arm, single center observational study to evaluate factors which were easily available from preoperative examination for predicting therapeutic effects and clinical prognosis of hepatic artery infusion chemotherapy (HAIC) for hepatocellular carcinoma. There factors are collected in preoperative routine blood examination, preoperative radiological imaging and pathological examination. Patients which are diagnosed with locally advanced hepatocellular carcinoma (HCC) will receive standard HAIC and follow-up exclusively as routinely done.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) remains a global health challenge and its incidence is growing worldwide. About 60%-70% of HCC patients were locally advanced or metastatic disease at the initial diagnosis, with a poor prognosis causing by unavailability of potentially curative therapies. Therefore, treatments that can control the progression and improve the prognosis of advanced HCC are under great need in sufficient liver reservation. Recent studies have shown that hepatic arterial infusion chemotherapy (HAIC) is beneficial to patients with locally advanced HCC. These studies have demonstrated that HAIC is superior to Sorafinib for the treatment of HCC with PVTT, whereas Sorafinib is recommended as first line treatment for locally advanced HCC. Therefore, HAIC is an important treatment option for locally advanced HCC. However, current tumor staging and prediction models for predicting the prognosis of HAIC for HCC is still unconvincing, and we found that some factors which were easily available from routine preoperative examination might be related to therapeutic effects and prognosis of HAIC for HCC. Thus, this prospective observational study aims to evaluate the value of these indicators for predicting therapeutic effects and prognosis of HAIC for HCC.

The standard procedure for HAIC is that femoral artery puncture and catheterization are performed in every cycle of treatment, a micro-catheter is inserted and located in feeding hepatic artery. The therapeutic scheme is modified FOLFOX6 regimens including oxaliplatin (130 mg/m2 infusion for 3 hours on day 1), leucovorin (200 mg/m2 from hour 3 to 5 on day 1) and Fluorouracil (400 mg/m2 in bolus, and then 2,400 mg/m2 continuous infusion 46 hours). All chemo-drugs are given by HAI. Treatment was repeated every 3 weeks and continued until intrahepatic lesions progression or unacceptable toxicity. Enhanced CT or MRI was performed every 6 weeks after treatment begins. Routine follow-up intervals were 2-4 months.

Before treatment, each patient will undergo routine hematological examinations which include blood routine, biochemical routine, coagulation routine, HCC related tumor markers. A three-phases enhanced CT or MR scan and biopsy of intrahepatic mass are performed before HAIC. Some factors through these examinations are collected and used to evaluate the relation of postoperative response rate and survival.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures.
* Cytohistological confirmation is required for diagnosis of HCC.
* Patients with advanced (unresectable and/or metastatic, stage C based on Barcelona-Clinic Liver Cancer [BCLC] staging classification) hepatocellular carcinoma which would not be suitable for treatment with loco-regional therapies or have progressed following locoregional therapy such as surgical resection, percutaneous hepatic arterial embolization, radiofrequency ablation, and percutaneous interventional therapy.
* At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1. Lesions previously treated with local therapy, such as radiation therapy, hepatic arterial embolization, radiofrequency ablation, and percutaneous interventional therapy should not be selected unless progression is noted at baseline, in which case, these lesions would be considered as non-target lesions.
* Current cirrhotic status of Child-Pugh class A-B, with no encephalopathy. Ascites controlled by diuretics is permitted in this study.
* Availability of a representative tumor tissue specimen (archival tumor tissue is allowed) at pre-screening.
* Eastern Cooperative Oncology Group Scale for Assessment of Patient Performance Status ≤ 2.
* Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial.
* Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to procedure:
* Hemoglobin > 100g/L
* Absolute neutrophil count >3.0 ×109/L
* Neutrophil count > 1.5 ×109/L
* Platelet count ≥ 50.0 ×109/L
* Total bilirubin < 51 μmol/L
* Alanine transaminase (ALT) and aminotransferase (AST) < 5 x upper limit of normal
* Albumin > 28 g/L
* Prothrombin time (PT)-international normalized ratio (INR) < 2.3, or PT < 6 seconds above control
* Serum creatinine < 110 μmol/L
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

* Received any prior systemic chemotherapy or molecular-targeted therapy for HCC such as sorafenib, lenvatinib.
* Previous local therapy completed less than 4 weeks prior to the dosing and, if present any related acute toxicity > grade 1.
* Any contraindications for hepatic arterial infusion procedure:
* Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).
* Renal failure / insufficiency requiring hemo-or peritoneal dialysis.
* Known severe atheromatosis.
* Known uncontrolled blood hypertension (> 160/100 mm/Hg).
* Patients with any other malignancies within the last 3 years before study start.
* History of HCC tumor rupture.
* Patients with severe encephalopathy.
* Patients with known active bleeding (e.g. from GI ulcers, esophageal varices) within 2 months prior to baseline/screening visit or with history or evidence of inherited bleeding diathesis or coagulopathy.
* Clinically significant (CTC grade 3 or 4) venous or arterial thrombotic disease within past 6 months.
* History of cardiac disease:
* Congestive heart failure >New York Heart Association (NYHA) class 2 (refer to Appendix 13.9).
* Active coronary artery disease (CAD) (myocardial infarction more than 6 months prior to study entry is allowed).
* Cardiac arrhythmias (>Grade 2 NCI-CTCAE Version 4.0) which are poorly controlled with anti-arrhythmic therapy or requiring pace maker.
* Uncontrolled blood hypertension (> 160/100 mm/Hg).
* Serious, non-healing wound, ulcer, or bone fracture.
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within past 6 months prior to study treatment.
* Clinically significant third space fluid accumulation (i.e., ascites requiring tapping despite use of diuretic or pleural effusion that either required tapping or is associated with shortness of breath).
* Patients who have undergone major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks of the start of protocol treatment.
* History of a bone marrow or solid organ transplant.
* Use of biologic response modifiers, such as G-colony stimulating factor (CSF), within 3 weeks prior to start of study drug. (G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however, they may not be substituted for a required dose reduction). Subjects taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 1 month prior to the study or during the study.
* Any other condition that would, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable or unwilling to swallow medication, social/ psychological issues, etc.
* Unable to undergo either contrast-enhanced magnetic resonance imaging (MRI) or contrast-enhanced computed tomography (CT).
* Known history of human immunodeficiency virus (HIV) seropositivity. HIV testing is not required as part of this study.
* Patients who have received any other investigational agents within a period of time that is less than the cycle length used for that treatment or equal to 4 weeks (whichever is shorter) prior to starting study drug and recovered from any side effects to grade 1 or less.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients which are diagnosed with locally advanced HCC will receive standard HAIC and follow-up exclusively as routinely done.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3-years Followed up
  Absence of death of any cause
Tumor Response | 3-years Followed up
  Tumor response to HAIC according to RECIST 1.1

SECONDARY OUTCOMES:
Progress Free Survival | 3-years Followed up
  Absence of disease progression other than death
Tumor local control | 3-years Followed up
  Absence of regrowth inside the treated lesion
Hepatic control | 3-years Followed up
  Absence of regrowth or onset of new lesions inside the liver
Distant control | 3-years Followed up
  Absence of extrahepatic progression

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, M.D., Principal Investigator — Department of Minimally Invasive and Interventional Radiology, Liver Cancer
Locations (1):
- Department of Minimally Invasive and Interventional Radiology, Liver Cancer Study and Service Group, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Background] Lyu N, Lin Y, Kong Y, Zhang Z, Liu L, Zheng L, Mu L, Wang J, Li X, Pan T, Xie Q, Liu Y, Lin A, Wu P, Zhao M. FOXAI: a phase II trial evaluating the efficacy and safety of hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin for advanced hepatocellular carcinoma. Gut. 2018 Feb;67(2):395-396. doi: 10.1136/gutjnl-2017-314138. Epub 2017 Jun 7. No abstract available. PMID 28592441